CLINICAL TRIAL: NCT02470715
Title: Identifying Molecular Drivers of Cancer
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: AMEM-2014-CCD001
Record Dates: First submitted 2015-06-09; First posted 2015-06-12 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Cancer; Tumor; Advanced Cancer
Keywords: genetic sequencing; genome; cancer; DNA; RNA; protein; metabolite
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Participants will have up to 3 blood tubes (about 30 ml) drawn under the condition that protocol criteria for blood sampling is met. Blood samples may be collected each time a participant undergoes a provider-ordered blood draw. Urine samples may also be collected approximately every 4-6 weeks.
  Participants may be asked to provide approximately 60-120 ml of first-morning-void urine. Tissue from a standard care surgical procedure or biopsy may be obtained. Additional core biopsies (for research) or excess surgical waste will be collected during each biopsy procedure when appropriate and will be processed and stored.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Molecular profile: Molecular profiled group receiving treatment based on genetics
  Interventions: Genetic: Molecular profile

INTERVENTIONS:
Genetic: Molecular profile — Patients and their treating physician will obtain the patient's genetic risk assessment
  Other Names: Genomic targeting

SUMMARY:
The primary aim of this study is to identify drivers of cancer by performing comprehensive genetic, proteomic, and metabolomic characterization of patient samples as a basis for understanding the underlying cause of disease.

DETAILED DESCRIPTION:
This study involves looking at the DNA, RNA, proteins, and metabolites in blood and tissue samples collected from subjects and linking them to their health information. By doing so, researchers hope to discover the underlying molecular causes of human diseases with the hope that this information can be used for the development of diagnostic tests and more effective treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnoses with cancer but healthy enough to undergo a biopsy procedure
* Between the ages of 18 and 100

Exclusion Criteria:

* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with cancer
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Genetic profiling | Up to 15 years
  To determine genetic changes associated with the development and growth of human disease. This should lead to better ways to detect, prevent, and treat a wide variety of human health conditions, including cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Leyland-Jones, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Cancer Institute, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Undecided